CLINICAL TRIAL: NCT07298109
Title: Investigating the Effectiveness of Diaphragmatic Release in Patients With Low Back Pain.
Brief Title: Diaphragmatic Release for Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Musa Güneş, Principal Investigator, PhD, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Low back pain-01
Record Dates: First submitted 2025-12-11; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain; Diaphragm; Relaxation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): In addition to spinal stabilization exercises, patients will undergo manual diaphragmatic release three times a week for eight weeks.
  Interventions: Other: Manual diaphragm release
- Control Group (Other): Patients in the control group will receive spinal stabilization exercises three times a week for eight weeks.
  Interventions: Other: Control

INTERVENTIONS:
Other: Manual diaphragm release — In addition to spinal stabilization exercises, patients will perform diaphragmatic relaxation exercises three days a week for eight weeks.
  Arms: Treatment Group
Other: Control — Patients will undergo spinal stabilization exercises three times a week for eight weeks.
  Arms: Control Group

SUMMARY:
Low back pain is one of the most common musculoskeletal disorders, significantly affecting the quality of life of individuals. In non-specific low back pain, a lack of stabilization in the core region negatively impacts the performance of activities. The diaphragm forms the framework of the core region, and its dysfunction can contribute to both respiratory problems and low back pain. This study will investigate the effects of diaphragm relaxation, added to spinal stabilization exercises, on pain, disability, quality of life, central sensitization, and trunk muscle endurance.

DETAILED DESCRIPTION:
Low back pain is one of the most common musculoskeletal problems, limiting daily life activities, leading to loss of productivity, and significantly reducing quality of life. In non-specific low back pain, insufficient stabilization in the trunk region and inadequate activation of deep muscles reduce the effectiveness of functional movements and contribute to chronic pain. The diaphragm, a crucial component of trunk stability, plays a critical role not only in respiratory function but also in maintaining spinal stability through the regulation of intra-abdominal pressure. Dysfunction or insufficient relaxation of the diaphragm can lead to changes in breathing patterns, impaired postural control, and persistent low back pain.

Therefore, a better understanding of the diaphragm's role in low back pain mechanisms and its targeting in therapeutic interventions is becoming increasingly important. This study aims to investigate the effects of diaphragm relaxation techniques, applied in addition to spinal stabilization exercises, on pain intensity, disability level, quality of life, central sensitivity, and trunk muscle endurance.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-65 years of age
* Having been diagnosed with chronic non-specific lower back pain (pain between the gluteal folds and the 12th ribs lasting at least 12 weeks and without a known pathoanatomical cause)
* Being willing to participate in the study

Exclusion Criteria:

* Psychological disorders, mental disorders, cancer, and severe depression
* History of primary or metastatic spinal malignancy or spinal fracture
* Neurological disease (Hemiplegia, Multiple Sclerosis, Parkinson's, etc.)
* Having been diagnosed with advanced osteoporosis
* Having undergone previous surgery or had an acute infection in the lumbar region

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Pain severity | Baseline, After intervention (eight week later)
  The severity of back pain will be assessed using the Visual Analog Scale (VAS). Patients choose the appropriate score between 0 and 10. Higher scores indicate higher pain levels.
Central sensitization | Baseline, After intervention (eight week later)
  Central sensitization will be assessed with the "Central Sensitization Scale". The total score range is between 0-100 points. As the score increases, sensitization increases and 40 points and above are considered higher sensitization.
Disability levels | Baseline, After intervention (eight week later)
  Disability will be measured by the Oswestry Disability Index. The total score ranges from 0-100 and the higher the score, the higher the level of disability.
Quality of life level | Baseline, After intervention (eight week later)
  In the SF-36 quality of life assessment, each sub-parameter is scored on a scale of 0. 0 is the lowest score and 100 is the highest.
Trunk muscle endurance | Baseline, After intervention (eight week later)
  The endurance of the trunk flexor and extensor muscles will be evaluated. Increasing the duration of the test indicates an increase in endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Musa Güneş, PhD, Principal Investigator — Karabuk University; Mustafa Kavak, PhD, Principal Investigator — Karabuk University; Aydın Sinan Apaydın, MD, Principal Investigator — Karabuk University
Locations (1):
- Karabuk University, Physiotherapy and Rehabilitation Application and Research Center, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No